CLINICAL TRIAL: NCT06888817
Title: Bevacizumab for the Treatment of Cerebral RAdiation Induced NecrosiS (BRAINS) Study: a Multicenter, Open-label, Randomized Clinical Trial to Assess the Clinical Efficacy and Cost-effectiveness of Bevacizumab Versus Corticosteroids as First-line Treatment in Patients With Symptomatic Cerebral Radiation Necrosis After Radiation for High-grade Glioma or Brain Metastases
Brief Title: Bevacizumab Versus Corticosteroids as First-line Treatment in Patients With Symptomatic Cerebral Radiation Necrosis After Radiation for High-grade Glioma or Brain Metastases
Acronym: BRAINS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UMC Utrecht (Other); Amsterdam UMC (Other); Medical Center Haaglanden (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23BNS
Record Dates: First submitted 2025-02-26; First posted 2025-03-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Radiation Necrosis; High Grade Glioma (III or IV); Brain Metastasases; Radiation Toxicity; Radiation Effect; Radiation Injury; Radiation Injuries
Keywords: Cerebral radiation necrosis; High Grade Glioma; Brain Metastases; Bevacizumab; Dexamethasone; Randomized Clinical Trial; First-line treatment; Anti-VEGF monocolonal antibody; Corticosteroids; Radiation induced necrosis; Radiation effects; Radiation injury; Radiation toxicity
MeSH Terms: conditions — Glioma; Radiation Injuries; Brain Neoplasms | interventions — Bevacizumab; Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bevacizumab (Experimental): Intravenous bevacizumab at a 600 mg flat dose every three weeks for four courses over 12 weeks
  Interventions: Drug: Bevacizumab; Drug: Dexamethasone
- Dexamethasone (Active Comparator): Daily oral dexamethasone followed by a protocol-based tapering dose over 12 weeks
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Bevacizumab — Intravenous bevacizumab at a 600 mg flat dose every three weeks for four courses over 12 weeks
  Other Names: Avastin; Anti-VEGF monoclonal antibody
  Arms: Bevacizumab
Drug: Dexamethasone — Daily oral dexamethasone followed by a protocol-based tapering dose over 12 weeks
  Other Names: Corticosteroids

SUMMARY:
Cerebral radiation necrosis (CRN) is a severe complication of high-dose radiation for brain metastases (BM) or glioma, which can potentially cause significant neurologic symptoms leading to serious morbidity and impaired quality of life (QoL). The first-line therapy for symptomatic CRN (sCRN) is corticosteroids, primarily dexamethasone, which often leads to complications, refractory symptoms, and interference with anti-cancer treatment. Since 2017, bevacizumab, an antibody against Vascular Endothelial Growth Factor (VEGF), has been used in a second-line treatment setting for refractory sCRN. A small randomized clinical trial (RCT) has shown that bevacizumab significantly diminishes cerebral edema on MRI and decreases clinical symptoms of sCRN in irradiated glioma patients. Several non-randomized clinical studies demonstrated a beneficial radiological and clinical effect of bevacizumab in patients with sCRN after irradiation for BM. The optimal first-line treatment for sCRN is currently unknown. Effective and safe first-line treatment of sCRN will optimize the patient's well-being and health-related QoL. Furthermore, minimizing corticosteroid use will benefit the clinical treatment options and outcomes of concomitant or future anti-cancer treatment. This phase III multicenter, open-label, randomized clinical trial compares the clinical efficacy of first-line bevacizumab versus standard-of-care dexamethasone for sCRN in patients with high-grade glioma (HGG) or BM.

DETAILED DESCRIPTION:
The primary objective of this trial is to compare the clinical efficacy of first-line bevacizumab versus dexamethasone for sCRN in HGG and BM patients at 12 weeks.

Both patients with HGG and patients with BM will be randomly assigned in a 1:1 ratio to one of two following treatment arms.

ARM 1 Intervention arm: intravenous bevacizumab at a 600 mg flat dose every three weeks for four courses over 12 weeks at hospital daycare.

ARM 2 Control arm: daily oral dexamethasone followed by a protocol-based tapering dose over 12 weeks.

Patients in the intervention (bevacizumab) arm may use dexamethasone concurrently with bevacizumab if clinically indicated.

The study treatment will be administered over 12 weeks, with a follow-up period of 2 years. Patients in both arms will have regular inpatient hospital visits and MRI brain scans, complete the Amsterdam Cognition scan twice during treatment, complete QoL, epilepsy, productivity, and medical costs questionnaires during treatment and follow up, and undergo optional blood withdrawal for translational research purposes. Standard of care laboratory blood tests during treatment depend on the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

Inclusion all patients (both HGG and BM):

1. Age ≥ 18 years old
2. First episode of sCRN ≥ 3 months after completion of focal (re-)irradiation, as determined by the local Multidisciplinary Neuro-Oncology Board. A clear working diagnosis of CRN without evidence of a combination with tumour progression is required
3. KPS score ≤ 90 and a minimum loss of two points in at least one domain of the NANO scale as compared to the maximum score of at that domain due to sCRN
4. Maximum daily dexamethasone use of 1 mg/day for the 8 weeks preceding randomization

   1. Dexamethasone may have been prescribed for various indications, except for managing (ongoing) cerebral edema
   2. Higher doses of dexamethasone are permitted during the week immediately preceding randomization if used specifically for the treatment of sCRN
5. Able to understand the patient information, online tests and questionnaires
6. Written informed consent

Inclusion BM:

1. BM of solid tumour, including all primary tumour types

Inclusion HGG:

1. A confirmed histological diagnosis of high-grade diffuse glioma according to WHO 2021 criteria, including: astrocytoma, IDH-mutant, grade 3-4; astrocytoma, IDH-wildtype (sybtype molecular glioblastoma); oligodendroglioma, 1p/19q codeleted, grade 3; diffuse glioma, NEC, grade 3-4; or glioblastoma, IDH-wildtype, grade 4

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study, both for the BM and HGG group:

1. Prior treatment with bevacizumab <6 months before diagnosis of sCRN
2. Life expectancy <3 months
3. Impending radiological or clinical signs of brain herniation necessitating immediate decompressive surgery
4. Any comorbidity or condition that prevents safe administration of the studied medication, determined by the treating physician, including but not limited to:

   1. Intolerance for murine proteins
   2. Hypersensitivity or allergy to the active substance or to any of the excipients of bevacizumab or dexamethasone
   3. Nephrotic syndrome or abnormal renal function

      o Calculated (Cockcroft-Gault) or measured creatinine clearance <30 mL/min; urine dipstick for proteinuria ≥ 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hours urine collection and must demonstrate ≤ 1 g of protein/24 hr.
   4. Clinical significant cardiovascular disease

      * Uncontrolled hypertension (systolic BP >150mmHg and/or diastolic >100mmHg) despite the use of ≥ 3 antihypertensive drugs
      * Previous hypertensive crisis, hypertensive encephalopathy or previous reversible posterior leukoencephalopathy syndrome (RPLS)
      * Non tumour related vascular event (e.g. cerebral or cardiac ischemia/bleeding (including transient ischemic attack, cerebral ischemia, unstable angina or angina requiring intervention, myocardial infarction), peripheral arterial thrombus, peripheral artery disease, deep venous thrombosis, lung embolism) < 6 months
      * History of aortic aneurysm or dissection
      * Congestive heart failure NYHA II-IV
   5. History of gastro-intestinal fistula, perforation or abscess < 6 months
   6. History of bleeding

      * Relevant pulmonary hemorrhage/ hemoptysis < 1 month or the presence of a pulmonary lesion with a high risk of bleeding (= central lung tumour and/or untreated squamous cell carcinoma) according to the treating physician
      * Active gastrointestinal bleeding < 6 months
      * Evidence of recent intracranial hemorrhage on MRI brain <3 months. Asymptomatic presence of hemosiderin depositions or punctate hemorrhage in the tumour do not serve as a ground for exclusion
   7. Excess risk of bleeding

      * History or evidence of inherited bleeding diathesis or significant coagulopathy with the risk of bleeding
      * Decreased platelet count < 75x109/L
   8. Risk of wound healing complications

      * Significant non-healing wound, (peptic) ulcer or bone fracture
      * Major surgical procedure (including open biopsy) or significant traumatic injury within 28 days prior to first study treatment or planned surgical procedure within the following next 28 days after planned study inclusion
      * Minor surgical procedure, stereotactic/core biopsy, fine needle aspiration within 7 days prior to first study treatment
   9. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hours urine collection and must demonstrate ≤ 1 g of protein/24 hr.
   10. Previous, current or planned high dose radiotherapy in the abdomen
   11. Pregnancy or lactation. Women of child bearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to randomization. WOCBP and female partners of male patients must comply with adequate contraception methods as requested by the study protocol
   12. Evidence of any other medical conditions (such as psychiatric illness, physical examination or laboratory findings) that may interfere with the study treatment, affect patient compliance or place the patient at high risk for treatment-related complications according to the treating physician
   13. Current or recent (within 30 days of first study treatment) treatment with another investigational drug or participation in another interventional study In case of uncertainty, consult the principal investigator of the study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy, defined as ≤ 1.5mg dexamethasone/day with one of the following 1) an improved KPS (of ≥ 10 points ) + at least stable NANO or 2) improved NANO (of ≥ 2 points) + at least stable KPS | 12 weeks
  The Karnofsky Performance Score (KPS) is a standard tool used to assess a patients' overall functional status and ability to carry out daily activities. The KPS is scored on a scale of 0 to 100, with higher scores indicating better physical function and lower scores indicating greater disability or dependence on others for care.
  The Neurologic Assessment in Neuro-Oncology (NANO) scale consists of 9 relevant neurologic domains (gait, strengths, ataxia, sensation, visual fields, facial strengths, language, level of consciousness, and behavior), which can be quantified based on direct observation and testing during routine clinical visits. Each domain is subdivided into 3 or 4 levels of function with a score of 0 indicating normal function, and a score of 2 or 3 indicating the most severe level of deficit for that domain. The maximum possible score on the NANO scale is 23, reflecting the highest level of impairment.

SECONDARY OUTCOMES:
Health-related quality of life using the EORTC-QLQ-C30 | up to 2 years
  The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30) is a validated tool designed to assess the overall health-related quality of life in cancer patients. It consists of 30 items measuring five functional scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, pain, and nausea/vomiting), a global health status/quality of life scale, and five single items evaluating additional symptoms (dyspnea, insomnia, appetite loss, constipation, and diarrhea) as well as perceived financial impact.
  Each item is scored on a 4-point Likert scale (1 = "Not at all" to 4 = "Very much"), except for the global quality of life domain, which is rated on a 7-point Likert scale. For functional and global quality of life scales, higher scores indicate better functioning and quality of life. For symptom scales and single items, higher scores reflect greater symptom burden and worse quality of life.
Health-related quality of life using EORTC-QLQ-BN20 | up to 2 years
  The EORTC QLQ-BN20 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Brain Neoplasm 20) is a brain cancer-specific module designed to assess the quality of life in brain cancer patients. It consists of 20 items, including seven symptom items (headaches, seizures, drowsiness, hair loss, itchy skin, leg weakness, and bladder control) and four multi-item scales (future uncertainty, visual disorder, motor dysfunction, and communication deficit). Each item is scored on a 4-point Likert scale (ranging from 1 = "Not at all" to 4 = "Very much"). The total score is converted to a 0-100 scale, with higher scores indicating a worse quality of life due to greater symptom burden.
Health-related quality of life using the QLQ-IADL-BN32 | up to 2 years
  The EORTC QLQ-IADL-BN32 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Instrumental Activities of Daily Living in Brain Neoplasms 32) is a validated questionnaire designed to assess the quality of life of brain tumor patients in relation to their ability to perform instrumental activities of daily living (IADL). It consists of five multi-item scales and two single-item scales, with each item scored on a 4-point Likert scale (ranging from 1 = "Not at all" to 4 = "Very much"). The total score is converted to a 0-100 scale, where higher scores indicate a greater impairment in IADL and worse quality of life.
Clinical efficacy using the KPS | up to 2 years
  The Karnofsky Performance Score (KPS) is a standard tool used to assess a patients' overall functional status and ability to carry out daily activities. The KPS is scored on a scale of 0 to 100, with higher scores indicating better physical function and lower scores indicating greater disability or dependence on others for care.
Clinical efficacy using the NANO scale | up to 2 years
  The Neurologic Assessment in Neuro-Oncology (NANO) scale consists of 9 relevant neurologic domains (gait, strengths, ataxia, sensation, visual fields, facial strengths, language, level of consciousness, and behavior), which can be quantified based on direct observation and testing during routine clinical visits. Each domain is subdivided into 3 or 4 levels of function with a score of 0 indicating normal function, and a score of 2 or 3 indicating the most severe level of deficit for that domain. The maximum possible score on the NANO scale is 23, reflecting the highest level of impairment.
Dexamethasone use | up to 2 years
  Dexamethasone tapering in mg/day
Clinical efficacy of 2 vs 4 cycles bevacizumab, with clinical efficacy defined as ≤ 1.5mg dexamethasone/day with one of the following 1) an improved KPS (of ≥ 10 points ) + at least stable NANO or 2) improved NANO (of ≥ 2 points) + at least stable KPS | 12 weeks
  The Karnofsky Performance Score (KPS) is a standard tool used to assess a patients' overall functional status and ability to carry out daily activities. The KPS is scored on a scale of 0 to 100, with higher scores indicating better physical function and lower scores indicating greater disability or dependence on others for care.
  The Neurologic Assessment in Neuro-Oncology (NANO) scale consists of 9 relevant neurologic domains (gait, strengths, ataxia, sensation, visual fields, facial strengths, language, level of consciousness, and behavior), which can be quantified based on direct observation and testing during routine clinical visits. Each domain is subdivided into 3 or 4 levels of function with a score of 0 indicating normal function, and a score of 2 or 3 indicating the most severe level of deficit for that domain. The maximum possible score on the NANO scale is 23, reflecting the highest level of impairment.
Cognitive functioning measured by the online cognitive test battery the Amsterdam Cognition Scan | 12 weeks
  Neurocognitive functioning will be assessed using the ACS (Amsterdam Cognition Scan) test battery at baseline and after 12 weeks. The ACS consists of seven online neuropsychological tests. Participants can complete the ACS remotely on their own computer at home, eliminating the need for an additional hospital visit. Each test within the ACS produces a standardized score, typically ranging from a minimum of 0 (indicating the lowest level of performance) to a maximum of 100 (indicating the highest level of performance). Higher scores reflect better cognitive functioning, while lower scores indicate greater cognitive impairment.
Radiologic response according to the RANO criteria | 12 weeks
  The Response Assessment in Neuro-Oncology 2.0 (RANO 2.0) criteria are an updated standardized framework for evaluating treatment response in patients with glioma. The Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria are used to evaluate treatment response in patients with brain metastases. A scoring system is not explicitly defined, but assessments are based on changes in contrast-enhancing and non-enhancing tumor components, as well as neurological status and corticosteroid dependency. Higher classifications indicating PD represent a worse outcome, signifying tumor growth or worsening symptoms.
  Lower classifications indicating CR or PR represent a better outcome, suggesting tumor reduction or stability.
Epileptic seizure control using the Seizure Control Composite Score Index | up to 2 years
  The Seizure Control Composite Score Index (SCCSI) is a standardized metric designed to assess seizure control by integrating both epileptic seizure frequency and antiseizure medication use. It provides a comprehensive evaluation of treatment effectiveness in reducing seizures while considering medication burden.
Treatment toxicity (CTCAE v5.0) | 15 weeks
  Incidence and severity of treatment toxicity of bevacizumab and dexamethasone according to CTCAE v5.0, reported for period of study treatment plus 21 days after. The percentage of patients reporting a grade 3 or higher, 4 or higher, or 5 at least possibly related to treatment will be reported.
Recurrence of symptomatic cerebral radiation necrosis | up to 2 years
  Recurrence of sCRN is defined as increase in edema volume on T2-weighted FLAIR images over that of the last MRI taken after treatment and necessity for treatment for recurrent sCRN (dexamethasone, bevacizumab, or surgery) due to neurological decline that is not attributable to tumour progression
Time to next symptomatic cerebral radiation necrosis treatment | up to 2 years
  Time to next sCRN treatment is defined as the time from completion of first-line dexamethasone/bevacizumab treatment for sCRN to initiating second-line treatment or reintroduction of treatment for sCRN
Tumour progression free survival | up to 2 years. After 2 years, yearly tumour progression (intra vs extra cranial) follow up will take place.
  Tumour progression free survival (PFS) is defined as the time from randomization to the first documented tumour progression as per RANO criteria for BM or HGG
Overall survival | up to 2 years. After 2 years, yearly survival follow up will take place.
  Overall survival (OS) is defined as time from randomization to death due to any cause
External validation prognostic tool | 1 year
  Validation of prognostic tool from retrospective BRAINS study for favourable clinical response (defined as in retrospective study: improvement of KPS by ≥ 10 points and dexamethasone tapering to ≤ 1.5 mg/day within 12 weeks following initiation of bevacizumab treatment) of second-line bevacizumab in first-line bevacizumab groups of the HGG and BM patient groups
Cost-effectiveness | 2 years
  Economic evaluation performing a cost-utility analysis (costs in relation to QALYs) from a societal perspective with a time horizon of two years for both HGG and BM patient groups

OTHER OUTCOMES:
Immuno-oncology protein biomarkers using Olink Target 96 Immuno-oncology panel | 12 weeks
  Immuno-oncology proteins as blood-based biomarkers for (early) treatment response in both treatment arms using Olink Target 96 Immuno-oncology panel
Tumour educated platelets | up to 2 years
  Platelet RNA profiles as blood-based biomarkers for (early) treatment response in both treatment arms
Pharmacokinetics bevacizumab and dexamethasone | 12 weeks
  Bevacizumab and dexamethasone serum and plasma concentrations pre- and post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dieta Brandsma, MD, PhD, Principal Investigator — Netherlands Cancer Institute - Antoni van Leeuwenhoek
Locations (5):
- Netherlands (5):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam
  - Amsterdam University Medical Centers, location VUmc and AMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Haaglanden Medical Center, The Hague
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No